CLINICAL TRIAL: NCT03783533
Title: Designing and Evaluating an Asynchronous Remote Communication Approach to Behavioral Activation With Clinicians and Adolescents At Risk for Depression
Brief Title: Adapting Behavioral Activation to Technology Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Jenness, Acting Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002824; P50MH115837 (NIH)
Record Dates: First submitted 2018-11-29; First posted 2018-12-21 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent Target Users of Behavioral Activation (BA) App (Experimental): Adolescents with PHQ-9 scores between 5 and 12 (Mild Range) who do not report current suicidality (Pine et al., 1999) will be recruited from clinician target users' practice settings. The investigators will recruit new adolescents for each Aim to decrease bias in feedback and outcomes.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Intervention: Behavioral Activation (BA) therapy is based on a functional analytic model of depression that highlights the need for increased positive reinforcement (rewards) and decreased anhedonia, or diminished motivation to seek rewards, to maintain normal mood. BA is significantly more effective than Cognitive Behavioral Therapy and comparable to antidepressant medication in reducing depressive symptoms among depressed adults (Dimidjian et al., 2006). McCauley (senior mentor) et al. (2016) adapted BA for adolescents to target anhedonia, effective problem solving and avoidant behaviors with peers, family, and school. McCauley's findings and others show BA is a promising intervention for adolescent MDD (Chu et al., 2009; Cuijpers et al.,, 2007; McCauley et al., 2015; Ritschel et al., 2011). BA focuses on targeting ideographically identified avoidant behaviors and rewarding experiences that affect mood.

SUMMARY:
This project aims to use an asynchronous remote communities (ARC) approach both to discover the design requirements for adapting Behavioral Activation (BA) to ARC as well as design/build an ARC platform for administering BA. The investigators will test the feasibility of our approach in a small feasibility observational study with clinicians and adolescents.

DETAILED DESCRIPTION:
An estimated 3.1 million adolescents are diagnosed with depression (MDD) each year (SAMHSA, 2016), and adolescent onset MDD is associated with chronic physical, mental and psychosocial disability (Birmaher et al., 1996). However, over 60% of adolescents with MDD do not receive mental health care, and, among those who do, treatment engagement is low (SAMHSA, 2016; Olfson et al., 2003). Behavioral Activation (BA) is an evidence-based psychosocial intervention (EBPI) for individuals with MDD (Dimidjian et al., 2006). While BA holds promise as an effective treatment with adolescents (McCauley et al., 2015, 2016), previous research approaches have found that adolescents may be better reached and engaged through social media, mobile technologies, and other technology platforms (Boyd, 2007; Park & Calamaro, 2013). In addition, BA requires frequent interaction from patients over time, which can be difficult and costly for clinicians to administer directly. Thus, there is an opportunity to improve usability and engagement of EBPIs via new technology-based tools. Asynchronous Remote Communities (ARC) is a promising technology-based approach for engaging adolescents that capitalizes on the reach of technology while also providing support, social interactions, and motivation to engage. ARCs are technology-mediated groups that use private online platforms to deliver weekly tasks to participants and gather information about perceptions in a format that is lightweight, accessible, usable, and low burden. The investigators aim to use ARC both to discover the design requirements for adapting BA to ARC as well as design/build an ARC platform for administering BA. The investigators will test the feasibility of our approach in a small feasibility study with clinicians and adolescents. The investigators propose the following specific aims:

Aim 1: Use the ARC approach with adolescents, primary care physicians, and mental health specialists to discover target user needs, design constraints and to observe their experience with ARC: The investigators will first use ARC to collect target user (i.e., primary care providers (PCP) and mental health specialists, adolescents at risk for depression) data to understand their needs and the facilitators and barriers to adapting BA to ARC.

Aim 2: Design & build an ARC platform for BA delivery with adolescents: Once the investigators have a strong understanding of the facilitators and barriers, the investigators will design a platform to use the ARC approach for BA delivery via Slack. The investigators will use an iterative design approach to understand the technical feasibility of the approach, whether and how to automate parts of the BA intervention using chatbots and other custom applications within Slack. The investigators will conduct small, informal usability testing with target users during this stage.

Aim 3: Test feasibility and usability with small pilot groups of adolescent and clinician target users: Once the investigators have a robust enough prototype of the ARC delivery platform for BA, the investigators will conduct a small pilot study with adolescents at-risk for depression and clinicians to assess the feasibility and usability of the approach. The investigators will collect data on the feasibility, usability, user burden, acceptability, and symptom outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with PHQ-9 scores between 5 and 15 (Mild to Moderate Range) who do not report current suicidality (Pine et al., 1999) will be recruited from clinician target users' practice settings.

Exclusion Criteria:

* Current suicidal ideation or PHQ-9 scores that are below or above the cutoff described above for adolescents.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To recruit teens between February and March 2020, we advertised our study in online groups, sent messages and flyers to clinicians, and a mailing list of parents with teenagers. Interested participants filled out a screener with contact information and the PHQ-8. If the teen was experiencing PHQ-8 >15, we required that they had a current therapist. Participants were paid $10 for each week's activity and $20 for exit interviews. All study activities were conducted between May and August 2020.
Groups:
- Adolescents: Adolescents with PHQ-9 scores between 5 and 20 who do not report current suicidality (Pine et al., 1999) will be recruited from clinician target users' practice settings. The investigators will recruit new adolescents for each Aim to decrease bias in feedback and outcomes.
  Behavioral Activation: Intervention: Behavioral Activation (BA) therapy is based on a functional analytic model of depression that highlights the need for increased positive reinforcement (rewards) and decreased anhedonia, or diminished motivation to seek rewards, to maintain normal mood. BA is significantly more effective than Cognitive Behavioral Therapy and comparable to antidepressant medication in reducing depressive symptoms among depressed adults (Dimidjian et al., 2006). McCauley (senior mentor) et al. (2016) adapted BA for adolescents to target anhedonia, effective problem solving and avoidant behaviors with peers, family, and school. McCauley's findings and others show BA is a promising intervention for adolescent MDD (Chu et al., 2009; Cuijpers et al.,, 2007; McCauley et al., 2015; Ritschel et al., 2011). BA focuses on targeting ideographically identified avoidant behaviors and rewarding experiences that affect mood.
Period: Overall Study
Arm/Group | Adolescents
Started | 11
Completed | 7
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Adolescents: Adolescents with PHQ-9 scores between 5 and 12 (Mild Range) who do not report current suicidality (Pine et al., 1999) will be recruited from clinician target users' practice settings. The investigators will recruit new adolescents for each Aim to decrease bias in feedback and outcomes.
  Behavioral Activation: Intervention: Behavioral Activation (BA) therapy is based on a functional analytic model of depression that highlights the need for increased positive reinforcement (rewards) and decreased anhedonia, or diminished motivation to seek rewards, to maintain normal mood. BA is significantly more effective than Cognitive Behavioral Therapy and comparable to antidepressant medication in reducing depressive symptoms among depressed adults (Dimidjian et al., 2006). McCauley (senior mentor) et al. (2016) adapted BA for adolescents to target anhedonia, effective problem solving and avoidant behaviors with peers, family, and school. McCauley's findings and others show BA is a promising intervention for adolescent MDD (Chu et al., 2009; Cuijpers et al.,, 2007; McCauley et al., 2015; Ritschel et al., 2011). BA focuses on targeting ideographically identified avoidant behaviors and rewarding experiences that affect mood.
Arm/Group | Adolescents
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.83 (2.14)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
  Non-binary/Transgender | 1
  Unknown | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Patient Health Questionnaire-8 [Mean (Standard Deviation); unit: units on a scale] — Measure of depression symptoms in the last 2 weeks. Scores range from 0 to 24 with higher scores indicating higher depression symptoms.
  units on a scale | 14.44 (3.94)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-Adolescent (PHQ-8)
Description: Measures symptoms of adolescent depression; Scores range from 0 to 24 with higher scores indicating higher depression symptoms.
Time Frame: Measured within 3-weeks post BA App User Testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescents
Number analyzed (Participants) | 5
units on a scale | 9.60 (6.27)

2. Primary Outcome: User Burden Scale
Description: Assesses the burden of the intervention adaptation with both clinician and adolescent participants across several domains and ranges from 0 to 80 for a total score with higher scores indicating higher burden. Scores were averaged across subscales including:
  * Access Burden
  * Emotional Burden
  * Financial Burden
  * Mental Burden
  * Physical Burden
  * Privacy Burden
  * Social Burden
  * Time Burden
Time Frame: Measured within 3-weeks post BA App User Testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescents
Number analyzed (Participants) | 5
units on a scale | .60 (.21)

3. Primary Outcome: Acceptability of Intervention Measure
Description: This is a survey measure that assesses the acceptability of the intervention adaptation with both clinician and adolescent participants. Scores range from 4 to 20 with higher scores indicating higher acceptability.
Time Frame: Measured within 3-weeks post BA App User Testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescents
Number analyzed (Participants) | 5
units on a scale | 3.55 (.51)

4. Primary Outcome: Appropriateness of Intervention Measure
Description: This is a survey measure that assesses the appropriateness of the intervention adaptation with both clinician and adolescent participants. Scores range from 4 to 20 with higher scores indicating higher appropriateness.
Time Frame: Measured within 3-week post BA App User Testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescents
Number analyzed (Participants) | 5
units on a scale | 3.4 (.55)

5. Primary Outcome: Feasibility of Intervention Measure
Description: This is a survey measure that assesses the feasibility of the intervention adaptation with both clinician and adolescent participants. Scores range from 4 to 20 with higher scores indicating higher feasibility.
Time Frame: Measured within 3-week post BA App User Testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescents
Number analyzed (Participants) | 5
units on a scale | 3.50 (.71)

6. Secondary Outcome: Platform Engagement
Description: Platform mood-activity logging across 35 days of possible logging 3x/day
Time Frame: Measuring platform engagement across 35 days of platform use.
Measure: Mean (Standard Deviation); unit: Number of mood-activity logs
Arm/Group | Adolescents
Number analyzed (Participants) | 5
Number of mood-activity logs | 52.13 (45.53)

ADVERSE EVENTS:
Time Frame: 4 months
Description: No differences in definition or additional information to provide
Arm/Group | Adolescents
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03783533/Prot_SAP_ICF_000.pdf